CLINICAL TRIAL: NCT04470973
Title: Population Pharmacokinetics of Amikacin and Cefuroxime in Critically Ill Septic Patients Admitted to the ICU or the ED
Brief Title: Pharmacokinetics of Amikacin and Cefuroxime in Critically Ill Patients.
Acronym: PHARAOH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PHARAOH
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Sepsis; Septic Shock; Infection, Bacterial; Critically Ill
Keywords: Sepsis; Septic Shock; Infection; Critically Ill
MeSH Terms: conditions — Sepsis; Shock, Septic; Bacterial Infections; Critical Illness; Infections | interventions — Cefuroxime; Amikacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and 24 hours urine will be collection following an intravenous gift of either cefuroxime or amikacin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cefuroxime/Amikacin: 20 patients will be included in the cefuroxime cohort and 20 patients in the amikacin cohort.
  Interventions: Drug: Cefuroxime; Drug: Amikacin

INTERVENTIONS:
Drug: Cefuroxime — Patients receive cefuroxime as part of standard care.
Drug: Amikacin — Patients receive amikacin as part of standard care.

SUMMARY:
Infections in critically ill patients are a major healthcare problem and an important source of morbidity and mortality. Since critically ill patients often have altered pharmacokinetics (PK) compared to non-critically ill patients there is a substantial risk that present standard dosing regimens of antibiotics lead to suboptimal outcomes for patients on the ICU or the ED. To prevent the risk of inadequate dosing in ICU patients, it is important to fully understand the PK of antibiotics in this vulnerable group in order to optimize the dosing regimens.

With this study, the investigators will describe the pharmacokinetics of cefuroxime and amikacin in ICU and ED patients. A heterogeneous population of ICU and ED patients will be included to be able to find which factors might influence the pharmacokinetics of these drugs and to what extent. By using population modeling the investigators will simulate different dosing regimens and MIC values and compare probability of target attainment between each of these dose and MIC combinations. This will allow the investigators to optimize dosing regimens of cefuroxime and amikacin in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is admitted to the ICU or ED;
2. The patient is at least 18 years of age on the day of inclusion;
3. Is managed with a central venous catheter or arterial line;
4. Is treated with amikacin and/or cefuroxime as standard care.

Exclusion Criteria:

1. Has previously participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to the ICU or ED.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
To describe the population pharmacokinetics of amikacin in Intensive Care or Emergency Department patients | 1 year
To describe the population pharmacokinetics of cefuroxime in Intensive Care or Emergency Department patients | 1 year

SECONDARY OUTCOMES:
To determine the influence of renal clearance and weight on the pharmacokinetics of amikacin and cefuroxime | 1 year
To determine the proportion of patients who attain adequate PK/PD targets in relation to the MIC of the suspected pathogen. | 1 year
To determine the toxicity of amikacin | 1 year

OTHER OUTCOMES:
To investigate to what extend renal replacement therapy affects the pharmacokinetics of amikacin and cefuroxime | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brüggemann, Phd, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc intensive care, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided